CLINICAL TRIAL: NCT02338466
Title: Randomized Therapeutic Study Assessing the Superiority of a Sequential Intravenous Thrombolysis Treatment (Rt-PA + Tenecteplase) in Comparison With Rt-PA Standard Treatment in Proximal Middle Cerebral Artery Occlusion (DIVA).
Brief Title: Superiority of Rt-PA + Tenecteplase in Comparison With Rt-PA Only in Proximal Middle Cerebral Artery Occlusion
Acronym: DIVA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Departure of the principal investigator and lack of succession
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13/EC/02
Record Dates: First submitted 2015-01-12; First posted 2015-01-14 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Nervous System Disorders; Cerebral Artery
MeSH Terms: conditions — Nervous System Diseases | interventions — Tissue Plasminogen Activator; Tenecteplase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rt-PA (Placebo Comparator): Patients treated by thrombolysis with rt -PA within 4h30 of the onset of symptoms to a proximal middle cerebral artery occlusion visible on a MRI 1 are pre- included. A second MRI ( IRM2 ) is performed between 1 hour and 1.5 hours after administration of rt-PA in the usual way .
  After the treatment by rt-PA, if there is no recanalization (TIMI score: 0,1, 2a), the patient is included. A patient included will be randomized either in the arm "rt-PA treatment only" or in the arm "rt-PA + tenecteplase treatment". If he is included in the arm "rt-PA only", he will not receive any other treatment for the study.
  Interventions: Drug: rt-PA
- rt-PA + tenecteplase (Active Comparator): If patient is in the arm "rt-PA + tenecteplase", he will receive tenecteplase (50UI/Kg) treatment. A third MRI will be performed at 24hour that will assess the recanalization status (TIMI), the final volume infarct and the hemorrhagic complications.
  Interventions: Drug: rt-PA; Drug: tenecteplase

INTERVENTIONS:
Drug: rt-PA — 0,9 mg/kg of rt-PA is infused intravenously 60 minutes, with 10% of the total dose administered as an initial intravenous bolus.
  Other Names: Actilyse
Drug: tenecteplase — Tenecteplase is under the form of powder and solvent for solution for injection.
  The maximum duration of this treatment is 15 seconds by a single bolus intravenous injection (0, 25 mg/kg).
  Other Names: Metalyse
  Arms: rt-PA + tenecteplase

SUMMARY:
Proximal Middle Cerebral Artery (MCA) occlusions constitute the most severe stroke. Intra-venous thrombolysis with rt-PA within the first 4,5 hours is the only proven effective treatment. Prognosis is closely related to the recanalization rate that reaches only 30 to 50%. A new therapeutic strategy consisting in a sequential intravenous (IV) thrombolysis by rt-PA followed by 50UI/kg of IV tenecteplase (TNK) has been proposed in case of no recanalization after rt-PA. A case series of 13 consecutive patients treated by this association has been published in 2011. A high rate of recanalization without hemorrhagic transformation increase has been reported. However, efficiency and safety of this therapeutic have to be assessed in a randomized multi-centric study. Such a study is of great interest since interventional neuroradiology has not already shown superiority regarding IV rt-PA. Moreover interventional neuroradiologists specialists are only available in major hospital and an IV sequential strategy could provide an interesting alternative.

Main study objectives:

Main Clinical Objective:

Sequential thrombolysis should be associated with a significant better outcome at 3-month, assessed by the modified Rankin score (mRS).

Main Radiological Objective:

Sequential thrombolysis should be associated with a higher rate of recanalization (TIMI 2b/3) at 24-hour.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, national, randomized, biomedical study comparing two therapeutic strategies in ischemic stroke associated with proximal middle cerebral artery occlusion.

Patients will be included in two randomized arms and the new sequential treatment approach (rt-PA + tenecteplase) will be compared with the standard treatment (rt-PA alone).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Cerebral infarction in relation with a proximal middle cerebral artery occlusion (M1 ou M2)
* NIHSS between 4 and 23
* Patient treated with intravenous rt-PA (0,9 mg/kg) within the first 4.5 hours
* No recanalization on the MRI performed 1 hour after rt-PA initiation (TIMI 0,1 ou 2a)
* Administration of TNK within the first 6 hours
* Informed and written consent obtained from the patient or next of kin
* Patient insured under the French social security system

Exclusion Criteria:

* Contraindication to MRI
* Contraindication to rt-PA administration
* Contraindication to TNK administration
* Contraindication to stroke thrombolysis
* Refusal to sign the informed consent
* Extensive small arteries disease (>5 microbleed and/or Fazekas score≥3)
* Systolic arterial pression> 185 mmHg or diastolic arterial pression > 110 mmHg
* Glycemia < 3 mmol/l (0,5g/l) or > 22 mmol/l (4g/l)
* Thrombopenia < 100 000/mm3 or INR > 1,5.
* Patients treated with new oral anticoagulant.
* Seizure as one of acute stroke symptoms
* Lumbar or arterial puncture in the previous 7 days or major surgery in the previous 15 days
* Carotid occlusion associated with MCA occlusion
* Thrombus length > 12mm assessed on gradient echo sequences
* Large DWI lesion, defined as ASPECTS < 7 / 10
* DWI/PWI Mismatch < 20% (when performed) on MRI 2
* Marked FLAIR hypersignal on cortical structure and light hypersignal on caudate or lenticular nucleus assessed on MRI 2.
* Parenchymal hemorrhage on MRI 2
* Pregnancy or breast feeding
* Patient currently included in a biomedical study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome ill be assessed at 3-month with the modified Rankin score by a blinded examiner. | 3 months
  The clinical outcome will be assessed at 3-month with the modified Rankin score by a blinded examiner.
  A score of 0-2 is considered good prognosis and a score 3-6 define a poor prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Julien JOUX, MD, Principal Investigator — Centre Hospitalier Universiatire de Martinique

IPD SHARING:
Plan to Share IPD: No